CLINICAL TRIAL: NCT01897441
Title: Prospective Tissue Collection in Breast Cancer Patients Receiving Preoperative Systemic Therapy
Brief Title: Chemotherapy Before Surgery and Tissue Sample Collection in Patients With Stage IIA-IIIC Breast Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interventional component of study terminated prior to full enrollment
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-02-079; NCI-2013-01194 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA013330 (NIH)
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Results first posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-11

CONDITIONS: Stage IIA Breast Cancer; Stage IIB Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Doxorubicin; Paclitaxel; Taxes; Trastuzumab; PF-05280014; Anastrozole; Letrozole; exemestane; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Stratum A: HER2-positive (Experimental): Patients receive Paclitaxel 80 mg/m^2 IV infusion over 1 hour for 12 weeks and Trastuzumab 8 mg/kg IV loading dose over 90 minutes, then 6 mg/kg IV every three weeks (after Paclitaxel when given concurrently) for a total of 17 doses over 51 weeks. Beginning 2-3 weeks after the last dose of Paclitaxel, patients receive Doxorubicin hydrochloride 60 mg/m^2 IV over 5-10 minutes and Cyclophosphamide 600 mg/m^2 IV infusion over 30-60 minutes every 2 weeks for 8 weeks.
  Interventions: Drug: Cyclophosphamide; Other: Cytology Specimen Collection Procedure; Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Biological: Trastuzumab
- Stratum B: HER2-negative (Experimental): Patients receive sequential Paclitaxel followed by Doxorubicin hydrochloride and Cyclophosphamide (AC) as described in Stratum A.
  Interventions: Drug: Cyclophosphamide; Other: Cytology Specimen Collection Procedure; Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel
- Stratum C: HER2-negative (Experimental): Patients receive sequential Doxorubicin hydrochloride and Cyclophosphamide (AC) followed by Paclitaxel. Patients receive Doxorubicin hydrochloride IV over 5-10 minutes and cyclophosphamide IV over 30-60 minutes every 2 weeks for 8 weeks. Patients then receive paclitaxel IV over 1 hour weekly for 12 weeks.
  Interventions: Drug: Cyclophosphamide; Other: Cytology Specimen Collection Procedure; Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel
- Stratum I: HER2-negative (Experimental): Patients receive Paclitaxel 80 mg/m^2 IV infusion over 1 hour for 12 weeks followed by Doxorubicin hydrochloride and Cyclophosphamide (AC). Patients receive Doxorubicin hydrochloride 60 mg/m^2 IV over 5-10 minutes and Cyclophosphamide 600 mg/m^2 IV infusion over 30-60 minutes every 2 weeks for 8 weeks.
  Interventions: Drug: Cyclophosphamide; Other: Cytology Specimen Collection Procedure; Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel
- Stratum II: HER2-positive (Experimental): Patients receive Paclitaxel 80 mg/m^2 IV infusion over 1 hour for 12 weeks and Trastuzumab 8 mg/kg IV loading dose over 90 minutes, then 6 mg/kg IV every three weeks (after Paclitaxel when given concurrently) for a total of 17 doses over 51 weeks. Beginning 2-3 weeks after the last dose of Paclitaxel, patients receive Doxorubicin hydrochloride 60 mg/m^2 IV over 5-10 minutes and Cyclophosphamide 600 mg/m^2 IV infusion over 30-60 minutes every 2 weeks for 8 weeks.
  Interventions: Drug: Cyclophosphamide; Other: Cytology Specimen Collection Procedure; Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Biological: Trastuzumab
- Stratum III: ER2-positive, HER2-negative (Experimental): Patients with ER-positive, HER2-negative disease may receive neoadjuvant endocrine therapy (NET) with an aromatase inhibitor: (either Anastrozole 1 mg po daily; Letrozole 2.5 mg po daily, Exemestane 25 mg po daily or Tamoxifen 20 mg po daily) for 4-6 months prior to surgery (or longer if clinically indicated). Anastrozole for 6 months is the preferred regimen for NET.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis; Drug: Endocrine therapy

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
  Arms: Stratum A: HER2-positive; Stratum B: HER2-negative; Stratum C: HER2-negative; Stratum I: HER2-negative; Stratum II: HER2-positive
Other: Cytology Specimen Collection Procedure — Correlative studies
  Other Names: Cytologic Sampling
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
  Arms: Stratum A: HER2-positive; Stratum B: HER2-negative; Stratum C: HER2-negative; Stratum I: HER2-negative; Stratum II: HER2-positive
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Stratum A: HER2-positive; Stratum B: HER2-negative; Stratum C: HER2-negative; Stratum I: HER2-negative; Stratum II: HER2-positive
Biological: Trastuzumab — Given IV
  Other Names: ABP 980; Anti-c-ERB-2; Anti-c-erbB2 Monoclonal Antibody; Anti-ERB-2; Anti-erbB-2; Anti-erbB2 Monoclonal Antibody; Anti-HER2/c-erbB2 Monoclonal Antibody; Anti-p185-HER2; c-erb-2 Monoclonal Antibody; HER2 Monoclonal Antibody; Herceptin; Herceptin Biosimilar PF-05280014; Herceptin Trastuzumab Biosimilar PF-05280014; MoAb HER2; Monoclonal Antibody c-erb-2; Monoclonal Antibody HER2; PF-05280014; rhuMAb HER2; Trastuzumab Biosimilar ABP 980; Trastuzumab Biosimilar PF-05280014
  Arms: Stratum A: HER2-positive; Stratum II: HER2-positive
Drug: Endocrine therapy — Patients with ER-positive, HER2-negative disease may receive neoadjuvant endocrine therapy (NET) with an aromatase inhibitor: (either Anastrozole 1 mg po daily; Letrozole 2.5 mg po daily, Exemestane 25 mg po daily or Tamoxifen 20 mg po daily) for 4-6 months prior to surgery (or longer if clinically indicated). Anastrozole for 6 months is the preferred regimen for NET.
  Other Names: Arimidex (anastrozole); Femara (letrozole); Aromasin (exemestane); Nolvadex (tamoxifen); Soltamox (tamoxifen)
  Arms: Stratum III: ER2-positive, HER2-negative

SUMMARY:
This pilot clinical trial studies chemotherapy before surgery and tissue sample collection in patients with stage IIA-IIIC breast cancer. Drugs used in chemotherapy, such as doxorubicin hydrochloride, cyclophosphamide, and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as trastuzumab, may interfere with the ability of tumor cells to grow and spread. Giving doxorubicin hydrochloride, cyclophosphamide, paclitaxel and trastuzumab may kill more tumor cells. Collecting and storing samples of tissue from patients with breast cancer to study in the laboratory may help doctors learn more about how well patients will respond to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the effects of preoperative neoadjuvant paclitaxel and doxorubicin (doxorubicin hydrochloride)/cyclophosphamide (AC) on: senescence; invasion/motility (tumor microenvironment of metastasis [TMEM] and 67 kDa laminin receptor [67LR]).

II. To create a biospecimen repository for future studies derived from patients with breast cancer receiving standard neoadjuvant chemotherapy.

OUTLINE: Patients with human epidermal growth factor receptor 2 (HER2)-positive disease are assigned to Stratum A, and patients with HER2-negative disease are randomized to Stratum B or C.

STRATUM A: Patients receive paclitaxel intravenously (IV) over 1 hour and trastuzumab IV over 30-90 minutes weekly for 12 weeks. Beginning 2-3 weeks later, patients receive doxorubicin hydrochloride IV over 5-10 minutes and cyclophosphamide IV over 30-60 minutes every 2 weeks for 8 weeks

STRATUM B: Patients receive paclitaxel, doxorubicin hydrochloride, and cyclophosphamide as in Stratum A.

STRATUM C: Patients receive doxorubicin hydrochloride IV over 5-10 minutes and cyclophosphamide IV over 30-60 minutes every 2 weeks for 8 weeks. Patients then receive paclitaxel IV over 1 hour weekly for 12 weeks.

Patients undergo surgery 2-6 weeks after the last chemotherapy dose.

In all arms, treatment continues in the absence of unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed adenocarcinoma of the breast associated with the following clinical stage: IIA, IIB, IIIA, IIIB, or IIIC; patients with stage IV disease are also eligible if there is an intention to perform breast surgery after neoadjuvant therapy is completed, or in patients participating in clinical trials where surgery after neoadjuvant therapy may be an option (eg. E2108)
* Estrogen receptor (ER), progesterone receptor (PR), and HER2/neu status documented by core needle biopsy of the primary tumor and/or regional lymph node must be known prior to beginning systemic therapy
* Patients must have had a bilateral diagnostic mammogram within 6 months of registration, and may also have a targeted sonography of the breast and/or ipsilateral axilla and magnetic resonance imaging (MRI) if clinically indicated
* Patients with clinically suspicious axillary lymph node involvement must have either aspiration cytology or biopsy prior to beginning therapy
* It is strongly encouraged that all patients have metallic clips placed in the tumor prior to neoadjuvant therapy in order to facilitate evaluation for microscopic disease at the time of surgery; placement of clips is particularly encouraged for patients being considered for breast conserving surgery
* No prior chemotherapy, irradiation, or definitive therapeutic surgery (eg, mastectomy or lumpectomy or axillary dissection) for this malignancy; patients who have had a prior sentinel lymph node biopsy for this malignancy are eligible
* Patients who received tamoxifen or another selective estrogen receptor modulator (SERM) for prevention or for other indications (e.g., osteoporosis, prior ductal carcinoma in situ [DCIS]) are eligible; tamoxifen therapy or other SERMs should be discontinued at least 1 week before the patient is enrolled on this study
* The patient is medically suitable candidate for preoperative chemotherapy and surgery in the judgment of the treating physicians
* Ability to understand and the willingness to sign a written informed consent document, and willing to provide blood samples before and during preoperative therapy; patients are also asked but not required to have research biopsies performed before and after therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-06; Primary Completion 2023-10-25 (Actual); Study Completion 2023-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Anampa, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

REFERENCES:
- [Background] Karagiannis GS, Pastoriza JM, Wang Y, Harney AS, Entenberg D, Pignatelli J, Sharma VP, Xue EA, Cheng E, D'Alfonso TM, Jones JG, Anampa J, Rohan TE, Sparano JA, Condeelis JS, Oktay MH. Neoadjuvant chemotherapy induces breast cancer metastasis through a TMEM-mediated mechanism. Sci Transl Med. 2017 Jul 5;9(397):eaan0026. doi: 10.1126/scitranslmed.aan0026. PMID 28679654

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 31 patients were enrolled into the study however one patient screen failed prior to being randomized into one of the study strata.
Groups:
- Stratum A: HER2-positive; Stratum II: HER2-positive: Patients receive Paclitaxel 80 mg/m^2 IV infusion over 1 hour for 12 weeks and Trastuzumab 8 mg/kg IV loading dose over 90 minutes, then 6 mg/kg IV every three weeks (after Paclitaxel when given concurrently) for a total of 17 doses over 51 weeks. Beginning 2-3 weeks after the last dose of Paclitaxel, patients receive Doxorubicin hydrochloride 60 mg/m^2 IV over 5-10 minutes and Cyclophosphamide 600 mg/m^2 IV infusion over 30-60 minutes every 2 weeks for 8 weeks.
  Cytology Specimen Collection Procedure:
  Correlative studies
  Laboratory Biomarker Analysis:
  Correlative studies
- Stratum B: HER2-negative: Patients receive sequential Paclitaxel followed by Doxorubicin hydrochloride and Cyclophosphamide (AC) as described in Stratum A.
  Cytology Specimen Collection Procedure:
  Correlative studies
  Laboratory Biomarker Analysis:
  Correlative studies
- Stratum C: HER2-negative: Patients receive sequential Doxorubicin hydrochloride and Cyclophosphamide (AC) followed by Paclitaxel. Patients receive Doxorubicin hydrochloride IV over 5-10 minutes and cyclophosphamide IV over 30-60 minutes every 2 weeks for 8 weeks. Patients then receive paclitaxel IV over 1 hour weekly for 12 weeks.
  Cytology Specimen Collection Procedure:
  Correlative studies
  Laboratory Biomarker Analysis:
  Correlative studies
- Stratum I: HER2-negative: Patients receive Paclitaxel 80 mg/m^2 IV infusion over 1 hour for 12 weeks followed by Doxorubicin hydrochloride and Cyclophosphamide (AC). Patients receive Doxorubicin hydrochloride 60 mg/m^2 IV over 5-10 minutes and Cyclophosphamide 600 mg/m^2 IV infusion over 30-60 minutes every 2 weeks for 8 weeks.
  Cytology Specimen Collection Procedure:
  Correlative studies
  Laboratory Biomarker Analysis:
  Correlative studies
- Stratum III: ER-Pos, HER2-negative: Patients with ER-positive, HER2-negative disease may receive neoadjuvant endocrine therapy (NET) with an aromatase inhibitor: (either Anastrozole 1 mg po daily; Letrozole 2.5 mg po daily, Exemestane 25 mg po daily or Tamoxifen 20 mg po daily) for 4-6 months prior to surgery (or longer if clinically indicated). Anastrozole for 6 months is the preferred regimen for NET.
  Cytology Specimen Collection Procedure:
  Correlative studies
  Laboratory Biomarker Analysis:
  Correlative studies
Period: Overall Study
Arm/Group | Stratum A: HER2-positive | Stratum B: HER2-negative | Stratum C: HER2-negative | Stratum I: HER2-negative | Stratum II: HER2-positive | Stratum III: ER-Pos, HER2-negative
Started | 1 | 8 | 9 | 5 | 6 | 1
Completed | 1 | 6 | 8 | 5 | 5 | 1
Not Completed | 0 | 2 | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawn by Provider | 0 | 2 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Stratum III: ER-positive, HER2-negative: Patients with ER-positive, HER2-negative disease may receive neoadjuvant endocrine therapy (NET) with an aromatase inhibitor: (either Anastrozole 1 mg po daily; Letrozole 2.5 mg po daily, Exemestane 25 mg po daily or Tamoxifen 20 mg po daily) for 4-6 months prior to surgery (or longer if clinically indicated). Anastrozole for 6 months is the preferred regimen for NET.
  Cytology Specimen Collection Procedure:
  Correlative studies
  Laboratory Biomarker Analysis:
  Correlative studies
- Total: Total of all reporting groups
Arm/Group | Stratum A: HER2-positive | Stratum B: HER2-negative | Stratum C: HER2-negative | Stratum I: HER2-negative | Stratum II: HER2-positive | Stratum III: ER-positive, HER2-negative | Total
Number analyzed (Participants) | 1 | 8 | 9 | 5 | 6 | 1 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 5 | 9 | 5 | 6 | 1 | 27
  >=65 years | 0 | 3 | 0 | 0 | 0 | 0 | 3
Age, Continuous [Mean (Full Range); unit: years] | 33 [33 to 33] | 52 [29 to 76] | 45 [26 to 60] | 56 [47 to 63] | 38 [29 to 48] | 56 [56 to 56] | 47 [26 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 8 | 9 | 4 | 6 | 1 | 29
  Male | 0 | 0 | 0 | 1 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 4 | 1 | 2 | 0 | 10
  Not Hispanic or Latino | 1 | 5 | 5 | 3 | 4 | 1 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 1 | 4 | 4 | 2 | 2 | 1 | 14
  White | 0 | 0 | 0 | 1 | 0 | 0 | 1
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 4 | 5 | 2 | 3 | 0 | 14
Region of Enrollment [Number; unit: participants]
  United States | 1 | 8 | 9 | 5 | 6 | 1 | 30

OUTCOME MEASURES:

1. Primary Outcome: Changes in Senescence and Secondary Biomarkers, Including TMEM, Mena, and 67LR
Description: Descriptive statistics by treatment group will be presented. The two-sampled t-test will be performed. Appropriate transformation may be used to improve normality of the outcome variable.
Time Frame: Baseline to 6 months
Population: Change in baseline to 6 month specimens for senescence, TMEM, mena, and 67LR biomarkers were not collected and analyzed.
Arm/Group | Stratum A: HER2-positive | Stratum B: HER2-negative | Stratum C: HER2-negative | Stratum I: HER2-negative | Stratum II: HER2-positive | Stratum III: ER-positive, HER2-negative
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Changes in Quantitative Biomarker Levels in Patients With Chemotherapy-responsive and -Resistant Tumors, Including Senescence, Cell Death, TMEM, Mena, and 67LR
Description: Paired T-test or Wilcoxon signed-rank test will be performed. Two-sample t-test will be performed to compare biomarker between the two groups. If the data are not normally distributed, a suitable data transformation such as the log or rank transformation will be applied. Logistic regression models will also be fit to the data with treatment sensitive/resistance category as the outcome and baseline as well as pre-post change in biomarker level as the main predictor variable to obtain estimates of odds ratios unadjusted and adjusted for potential confounders including patients characteristics.
Time Frame: Baseline to 8 weeks (2 courses)
Population: Change in baseline to 8 week specimens for cell death, TMEM, mena, and 67LR biomarkers were not collected and analyzed.
Arm/Group | Stratum A: HER2-positive | Stratum B: HER2-negative | Stratum C: HER2-negative | Stratum I: HER2-negative | Stratum II: HER2-positive | Stratum III: ER-positive, HER2-negative
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected up to 2-3 weeks post-treatment initiation in conjunction with biopsy collections, up to an overall period of 6-8 weeks total.
Description: In accordance with the study protocol only adverse events data related to the biopsy were considered research-related and were identified for collection and reporting as part of the clinical study.
Arm/Group | Stratum A: HER2-positive | Stratum B: HER2-negative | Stratum C: HER2-negative | Stratum I: HER2-negative | Stratum II: HER2-positive | Stratum III: ER-positive, HER2-negative
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/8 | 0/9 | 0/5 | 0/6 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/8 | 0/9 | 0/5 | 0/6 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/8 | 0/9 | 0/5 | 0/6 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-11): https://cdn.clinicaltrials.gov/large-docs/41/NCT01897441/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-25): https://cdn.clinicaltrials.gov/large-docs/41/NCT01897441/ICF_001.pdf